CLINICAL TRIAL: NCT01682915
Title: Structural and Functional Connectivity of Frontostriatal and Frontoparietal Networks as Endophenotypes of Attention-deficit Hyperactivity Disorder
Brief Title: Structural and Functional Connectivity of Frontostriatal and Frontoparietal Networks as Endophenotypes of ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Susan Shur-Fen Gau, National Taiwan University Hospital
Other Study IDs: 201204071RIC
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD; endophenotype; executive function; diffusion spectrum imaging; resting-state fMRI; frontostriatal and frontoparietal circuitries; DAT1
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Group 1: ADHD+DAT1, Probands: 30 ADHD probands with DAT1 variants
- Group 2: ADHD+DAT1, Unaffected sibling: 30 same-sex unaffected siblings of Group 1
- Group 3: ADHD Drug-naïve, Probands: 30 ADHD probands without DAT1 gene variants, who were age-, sex-, and IQ-matched to Group 1
- Group 4: ADHD Drug-naïve, unaffected sibling: 30 same-sex unaffected siblings of Group 3
- Matched controls: 30 age-, sex- and IQ-matched TD controls for each of 4 groups

SUMMARY:
Attention deficit/hyperactivity disorder (ADHD) is a common, impairing, clinically and genetically heterogeneous neuropsychiatric disorder with lifelong executive dysfunctions. The ultimate goal of this 3-year case-control imaging genomic study with unaffected siblings and typically developing (TD) children as controls is to identify useful imaging endophenotype for ADHD by investigating the structural connectivity, as assessed by diffusion spectrum imaging (DSI), and functional connectivity, as assessed by resting-state fMRI (rsfMRI) of brain regions related to cognitive/executive controls with regards to the ADHD status and the presence of dopamine transporter gene variants (DAT1).

Specific Aims:

1. to validate the executive functions, visuospatial memory, and structural and functional connectivity in frontostriatal, and frontoparietal circuitries as effective neurocognitive endophenotypes;
2. to correlate the data from structural and functional connectivity, neuropsychology, and ADHD core symptoms stratifying by the presence of ADHD, proband-unaffected sibling dyads, and the presence of DAT1 variant; and
3. To investigate reported candidate genes, in addition to DAT1 variant, related to dopamine and noradrenergic neurotransmitter systems in the association with neurocognitive endophenotypes such as DRD1, DRD2, DRD4, DRD5, DBH, MAO-A, ADRA2A, ADRA2C, NET, and COMT.

DETAILED DESCRIPTION:
The sample (n=240, 8 groups, ages 10-20, IQ > 80) consists of (1) 30 ADHD probands with DAT1 variants, (2) 30 same-sex unaffected siblings, (3) 30 ADHD probands without DAT1 gene variants, who were age-, sex-, and IQ-matched to Group 1, (4) 30 same-sex unaffected siblings of Group 3, (5) 30 age-, sex- and IQ-matched TD controls for each of 4 groups (Groups 1, 2, 3 & 4).

The assessments include psychiatric interviews, self-administered questionnaires (CBCL and SNAP-IV for ADHD and behavioral problems; the SAICA for school and social function), neurocognitive assessments (WISC-III-R or WAIS-III for intelligence, Conner's CPT for sustained attention, inhibition, and vigilance, CANTAB for executive functions and visuo-spatial memory), and MRI assessments (Structural MRI, DSI and rsfMRI).

Brain Imaging: (1) Structural MRI (T1- and T2-weighted images), DSI and rsfMRI data will be acquired on a 3T MRI system with a 32-channel head coil. DSI employs a pulsed-gradient spin-echo echo planar imaging (EPI) sequence by applying 102 diffusion gradient vectors and the maximum diffusion sensitivity = 4000 s/mm2, and rsfMRI is a 6-minute scan using a gradient-echo EPI sequence with 180 volumes. (2) Structural connectivity analysis: DSI tractography will be performed using in-house software (DSI studio, http://dsi-studio.labsolver.org/Home). Tracts-of-interest in the frontostriatal circuit and the frontoparietal circuit will be identified, and tract-specific analysis will be used to analyze the microstructural integrity along individual tract bundles. (3) Functional connectivity analysis: SPM8 program and in-house MATLAB codes will be used for analyses of rsfMRI data. Region-of-interests (ROIs) will be placed in the nodes of the corresponding circuits according to an anatomical template (WFU_PickAtlas 3.03). These ROIs will serve for tract determination in the tractography procedure and for seed regions in which BOLD signals are extracted for regression analysis among nodes.

ELIGIBILITY:
Inclusion Criteria:

* ADHD+DAT1 groups: Subjects aged 12-20, who have clinical diagnosis of ADHD according to the DSM-IV diagnostic criteria and who have risk alleles of DAT1 gene, regardless of having same-sex unaffected siblings or the drug-naïve status.
* ADHD drug-naïve groups: Subjects aged 12-20, who have clinical diagnosis of ADHD according to the DSM-IV diagnostic criteria, who do not have risk alleles of DAT1 gene, who have the same-sex unaffected siblings and who have never been treated by medication for treating ADHD.

Exclusion Criteria:

* These subjects will be excluded from the study if they have any of the following criteria: (1) Comorbidity with DSM-IV-TR diagnosis of pervasive developmental disorder, schizophrenia, schizoaffective disorder, delusional disorder, other psychotic disorder, organic psychosis, schizotypal personality disorder, bipolar disorder, depression, severe anxiety disorders or substance use; (2) With neurodegenerative disorder, epilepsy, involuntary movement disorder, congenital metabolic disorder, brain tumor, history of severe head trauma, and history of craniotomy; (3)With visual or hearing impairments, or motor disability which may influence the process of MRI assessment; and (4) Full-scale IQ lower than 80. In addition, if the control subjects have ODD or CD, they will be excluded.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample (n=240, 8 groups, ages 10-20, IQ > 80) consists of (1) 30 ADHD probands with DAT1 variants, (2) 30 same-sex unaffected siblings, (3) 30 ADHD probands without DAT1 gene variants, who were age-, sex-, and IQ-matched to Group 1, (4) 30 same-sex unaffected siblings of Group 3, (5) 30 age-, sex- and IQ-matched TD controls for each of 4 groups (Groups 1, 2, 3 & 4).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin HY, Kessler D, Tseng WI, Gau SS. Increased Functional Segregation Related to the Salience Network in Unaffected Siblings of Youths With Attention-Deficit/Hyperactivity Disorder. J Am Acad Child Adolesc Psychiatry. 2021 Jan;60(1):152-165. doi: 10.1016/j.jaac.2019.11.012. Epub 2019 Nov 26. PMID 31778781
- [Derived] Chiang HL, Hsu YC, Shang CY, Tseng WI, Gau SS. White matter endophenotype candidates for ADHD: a diffusion imaging tractography study with sibling design. Psychol Med. 2020 May;50(7):1203-1213. doi: 10.1017/S0033291719001120. Epub 2019 May 22. PMID 31115278